CLINICAL TRIAL: NCT02720653
Title: Determinants of Olfactory Dysfunction in Chronic Rhinosinusitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Dr. Timothy L. Smith, Professor, Chief of Rhinology, Oregon Health and Science University
Other Study IDs: DC005805-11
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chronic Rhinosinusitis; Olfactory Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mucus specimens will be collected and analyzed for cytokine profiles and proteomics
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Appropriate Medical Therapy: Patients will self-select continued, non-standardized, appropriate medical management of symptoms associated with chronic sinusitis.
- Endoscopic Sinus Surgery: Patients will self-select endoscopic sinus surgery for symptoms associated with chronic sinusitis.
  Interventions: Procedure: Endoscopic sinus surgery

INTERVENTIONS:
Procedure: Endoscopic sinus surgery
  Other Names: Sinus surgery
  Groups: Endoscopic Sinus Surgery

SUMMARY:
Olfactory dysfunction is a cardinal symptom of chronic rhinosinusitis, a disease which affects 12.5% of the adult population across all racial and ethnic groups. Previous research has documented olfactory deficit in 68% of patients with chronic rhinosinusitis and 20% with complete anosmia, suggesting that olfactory dysfunction affects over 25 million individuals in the United States with chronic rhinosinusitis. This proposed investigation will be used to predict olfactory outcomes following treatments for chronic rhinosinusitis and gain insights into mechanisms of olfactory dysfunction in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years of age)
* A diagnosis of medical recalcitrant CRS as defined by 2015 Adult Sinusitis Guidelines outlined by the American Academy of Otolaryngology
* Provide written informed consent and authorization.
* Study participants must be able to complete consent, all study evaluations, olfactory testing, and study-related health questionnaires written in the English language.
* Patients must self-select subsequent treatment option (endoscopic sinus surgery or continued medical therapy) to be dictated by the disease process and judgment and preferences of each individual, following counseling for each treatment option.
* Present to the enrolling site with indication for a CT scan or a CT scan completed, off-site, from another provider
* Complete appropriate standardized medical treatment by the Interim Assessment, 6-week follow-up period including, but not limited to, at least one course of either topical corticosteroids (>21-days) or a 5-day course of oral corticosteroid therapy, and at least one course (>14-days) of culture-directed or broad spectrum antibiotic therapy.

Exclusion Criteria:

* Children (< 18 years of age)
* Any patient unable and/or unwilling to complete questionnaires or clinical testing or cooperate with all study protocols.
* Non-English speaking / English translation services required
* Unwilling or unable to provide informed, written consent.
* Contra-indications for any type of continued medical therapy required for treatment of symptoms related to CRS
* Patients who have not undergone previous prescribed medical therapy as described in Inclusion Criteria.
* Individuals of any vulnerable population including: children, pregnant women, neonates, decisionally impaired adults, or prisoners.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present in clinic with indications of medically refractory chronic sinusitis.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Sniffin' Stick olfactory testing | 6 months
  Improvement in olfactory function

SECONDARY OUTCOMES:
22-Item Sinonasal Outcome Test | 6 months
  Improvement in disease specific quality of life
Questionnaire for Olfactory Dysfunction, QOD-NS | 6 months
  Improvement in olfactory specific quality of life

REFERENCES:
- [Derived] Tullis B, Mace JC, Massey C, Batterman S, Ramakrishnan VR, Beswick DM, Soler ZM, Smith TL, Alt JA, Gill AS. Pollen Exposure and Chronic Rhinosinusitis Quality of Life Disease Severity. Laryngoscope Investig Otolaryngol. 2025 Nov 13;10(6):e70309. doi: 10.1002/lio2.70309. eCollection 2025 Dec. PMID 41246125
- [Derived] Patel PA, Kallenberger EM, Nguyen SA, Mace JC, Duffy AN, Soler ZM, Smith TL, Schlosser RJ. Factors Affecting Nasal Discharge in Chronic Rhinosinusitis Patients. Laryngoscope. 2025 Nov;135(11):4086-4092. doi: 10.1002/lary.32288. Epub 2025 May 26. PMID 40417805
- [Derived] Pandrangi VC, Mace JC, Kim JH, Geltzeiler M, Detwiller KY, Soler ZM, Schlosser RJ, Alt JA, Ramakrishnan VR, Mattos JL, Smith TL. Work productivity and activity impairment in patients with chronic rhinosinusitis undergoing endoscopic sinus surgery-A prospective, multi-institutional study. Int Forum Allergy Rhinol. 2023 Mar;13(3):216-229. doi: 10.1002/alr.23070. Epub 2022 Aug 23. PMID 35938699
- [Derived] Gill AS, Beswick DM, Mace JC, Menjivar D, Ashby S, Rimmer RA, Ramakrishnan VR, Soler ZM, Alt JA. Evaluating Distance Bias in Chronic Rhinosinusitis Outcomes. JAMA Otolaryngol Head Neck Surg. 2022 Jun 1;148(6):507-514. doi: 10.1001/jamaoto.2022.0268. PMID 35511170
- [Derived] Allensworth JJ, Schlosser RJ, Smith TL, Mace JC, Soler ZM. Use of the Diet History Questionnaire III to determine the impact of dysosmia on dietary quality. Int Forum Allergy Rhinol. 2022 Jun;12(6):849-858. doi: 10.1002/alr.22926. Epub 2021 Dec 18. PMID 34762776
- [Derived] Soler ZM, Schlosser RJ, Bodner TE, Alt JA, Ramakrishnan VR, Mattos JL, Mulligan JK, Mace JC, Smith TL. Endotyping chronic rhinosinusitis based on olfactory cleft mucus biomarkers. J Allergy Clin Immunol. 2021 May;147(5):1732-1741.e1. doi: 10.1016/j.jaci.2021.01.021. Epub 2021 Feb 4. PMID 33549569
- [Derived] Beswick DM, Smith TL, Mace JC, Alt JA, Farrell NF, Ramakrishnan VR, Schlosser RJ, Soler ZM. Ethmoid-to-maxillary opacification ratio: a predictor of postoperative olfaction and outcomes in nasal polyposis? Int Forum Allergy Rhinol. 2021 Jan;11(1):48-57. doi: 10.1002/alr.22625. Epub 2020 Jun 18. PMID 32558260
- [Derived] Thomas AJ, Mace JC, Ramakrishnan VR, Alt JA, Mattos JL, Schlosser RJ, Soler ZM, Smith TL. Quality-of-life and olfaction changes observed with short-term medical management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2020 May;10(5):656-664. doi: 10.1002/alr.22532. Epub 2020 Feb 3. PMID 32017433
- [Derived] Beswick DM, Ayoub NF, Mace JC, Mowery A, Hwang PH, Smith TL. Acute Exacerbations in Recurrent Acute Rhinosinusitis: Differences in Quality of Life and Endoscopy. Laryngoscope. 2020 Dec;130(12):E736-E741. doi: 10.1002/lary.28460. Epub 2019 Dec 14. PMID 31837149
- [Derived] Loftus C, Schlosser RJ, Smith TL, Alt JA, Ramakrishnan VR, Mattos JL, Mappus E, Storck K, Yoo F, Soler ZM. Olfactory cleft and sinus opacification differentially impact olfaction in chronic rhinosinusitis. Laryngoscope. 2020 Oct;130(10):2311-2318. doi: 10.1002/lary.28332. Epub 2019 Oct 11. PMID 31603563
- [Derived] Beswick DM, Mace JC, Soler ZM, Rudmik L, Alt JA, Smith KA, Detwiller KY, Ramakrishnan VR, Smith TL. Socioeconomic status impacts postoperative productivity loss and health utility changes in refractory chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Sep;9(9):1000-1009. doi: 10.1002/alr.22374. Epub 2019 Jun 27. PMID 31246360
- [Derived] Smith TL, Schlosser RJ, Mace JC, Alt JA, Beswick DM, DeConde AS, Detwiller KY, Mattos JL, Soler ZM. Long-term outcomes of endoscopic sinus surgery in the management of adult chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Aug;9(8):831-841. doi: 10.1002/alr.22369. Epub 2019 Jun 17. PMID 31207172
- [Derived] Alt JA, Orlandi RR, Mace JC, Soler ZM, Smith TL. Does Delaying Endoscopic Sinus Surgery Adversely Impact Quality-of-Life Outcomes? Laryngoscope. 2019 Feb;129(2):303-311. doi: 10.1002/lary.27473. Epub 2018 Sep 12. PMID 30208208
- [Derived] Beswick DM, Mace JC, Rudmik L, Soler ZM, DeConde AS, Smith TL. Productivity changes following medical and surgical treatment of chronic rhinosinusitis by symptom domain. Int Forum Allergy Rhinol. 2018 Dec;8(12):1395-1405. doi: 10.1002/alr.22191. Epub 2018 Jul 28. PMID 30054977
- [Derived] Beswick DM, Mace JC, Soler ZM, Ayoub NF, Rudmik L, DeConde AS, Smith TL. Appropriateness criteria predict outcomes for sinus surgery and may aid in future patient selection. Laryngoscope. 2018 Nov;128(11):2448-2454. doi: 10.1002/lary.27227. Epub 2018 May 14. PMID 29756211
- [Derived] Mattos JL, Schlosser RJ, Mace JC, Smith TL, Soler ZM. Establishing the minimal clinically important difference for the Questionnaire of Olfactory Disorders. Int Forum Allergy Rhinol. 2018 Sep;8(9):1041-1046. doi: 10.1002/alr.22135. Epub 2018 May 2. PMID 29719139
- [Derived] Othieno F, Schlosser RJ, Rowan NR, Storck KA, Mattos JL, Smith TL, Soler ZM. Taste impairment in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2018 Jul;8(7):783-789. doi: 10.1002/alr.22113. Epub 2018 Mar 23. PMID 29569385
- [Derived] Smith TL. THE 2017 13TH ANNUAL DAVID W. KENNEDY, MD, LECTURE The evolution of outcomes in sinus surgery for chronic rhinosinusitis: past, present, and future. Int Forum Allergy Rhinol. 2017 Dec;7(12):1121-1126. doi: 10.1002/alr.22026. Epub 2017 Oct 13. PMID 29028274
- [Derived] Beswick DM, Mace JC, Chowdhury NI, Alt JA, Hwang PH, DeConde AS, Smith TL. Comparison of surgical outcomes between patients with unilateral and bilateral chronic rhinosinusitis. Int Forum Allergy Rhinol. 2017 Dec;7(12):1162-1169. doi: 10.1002/alr.22020. Epub 2017 Sep 22. PMID 28941136
- [Derived] DeConde AS, Mace JC, Ramakrishnan VR, Alt JA, Smith TL. Analysis of factors associated with electing endoscopic sinus surgery. Laryngoscope. 2018 Feb;128(2):304-310. doi: 10.1002/lary.26788. Epub 2017 Aug 4. PMID 28776718